CLINICAL TRIAL: NCT03702478
Title: Quality of Life in Patients With and Without a Parastomal Bulge - a Cross-sectional Study of Patients in the Danish Stoma Database Capital Region
Brief Title: Quality of Life in Patients With and Without a Parastomal Bulge
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Novo Nordic Foundation (Other); Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Thordis Thomsen, Associate professor, Rigshospitalet, Denmark
Other Study IDs: 16021425
Record Dates: First submitted 2018-08-10; First posted 2018-10-11 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Quality of Life; Parastomal Hernia
Keywords: Quality of life; hernia; parastomal bulging; stoma; cross-sectional
MeSH Terms: conditions — Hernia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No intervention, cross-sectional study: Questionnaire, cross-sectional study
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — No intervention only observational

SUMMARY:
It is not well-established whether a parastomal bulge impacts stoma patients HRQoL or if HRQOL differs according to the underlying disease or type of stoma. In this large cross-sectinal study stoma patients with and without a parastomal bulge are asked about their health-related quality of life and stomarelated quality of life. Stoma patients are identified in the danish stoma database and contacted two times by email. Non-responders are sent a paper booklet.

DETAILED DESCRIPTION:
A cross-sectional study of patients registered in the Danish Stoma Database Capital Region (DSDCR), with permanent or temporary enterostoma after surgery performed between 2011 and 2016. Via a unique personal identification number registered in DSDCR patients will be contacted by e-mail using the e-Boks system, an official electronic distribution system covering around 80% of the Danish adult population. The e-mail will contain information about the study and a personal link to SurveyXact, an online survey program allowing for direct electronic data entry by patients. First reminder will be sent after one week and a second reminder again one week later. If necessary, a third reminder additionally three weeks later will be sent to patients by post, including a paper booklet of the questionnaires as described below.

For patients without e-Boks, DSDCR will be linked to the Danish Civil Registration System via the unique personal identification number, providing information on patient's addresses. Information on the study and a paper booklet of questionnaires will be sent to patients by post. A reminder will be sent by post after three weeks if necessary. Hereafter, no further attempts will be made to contact the patients. To include other relevant variables in the analysis of data, data from the Danish Anaesthesia Database (DAD) and the Danish Colorectal Cancer Database will be linked. Quality of life will be assessed using StomaQol and SF-36. Colostomy Impact score will also be obtained. Patients will self-report a parastomal bulge and information such as education, alcohol consumption, physical activity and civil status.

ELIGIBILITY:
Inclusion Criteria:

* permanent active sigmoideostomy, transverseostomy, jejunostomi or ileostomy
* temporary active sigmoideostomy, transverseostomy, jejunostomi or ileostomy

Exclusion Criteria:

* age younger than 18 years
* stoma closure at follow-up
* death

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients registered in the Danish Stoma Database Capital Region, having undergone stoma surgery between 2011 till end of 2016.
Sampling Method: Non-Probability Sample
Enrollment: 1453 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Health related quality of life (SF-36 ) and Stoma related Qol (StomaQol) in relation to stoma type or underlying condition | Up to 7 years after stoma formation
  Investigate and compare HRQoL in patients with and without a self-reported parastomal bulge in relation to an ileostomy or colostomy. HRQol is measured with SF-36 and StomaQol

SECONDARY OUTCOMES:
Exploration of the frequency of self-reported parastomal bulging | Up to 7 years after stoma formation
  Investigate the frequency of parastomal bulging
Relationship between symptoms and HRQOL measured with StomaQol | Up to 7 years after stoma formation
  Investigate the relationship between symptoms in the Stomaqol scale and overall score
Relationship between PB duration and HRQOL measured with StomaQol and SF-36 | Up to 7 years after stoma formation
  The association between duration of PB and overall scores on SF-36 and StomaQol
Relationship between PB size and HRQOL measured with SF-36 and StomaQol | Up to 7 years after stoma formation
  The association between duration of PB and overall scores on SF-36 and StomaQol

OTHER OUTCOMES:
Alcohol consumption measured by Time-line-follow-back | Up to 7 years after stoma formation
  Exploration of the distribution of alcohol consumption in stoma patients with and without parastomal bulging.
Physical activity measured with high or low intensity questions. A non-validated physical activity scale | Up to 7 years after stoma formation.
  Exploration of the distribution of high and low intensity physical activity in stoma patients with and without parastomal bulging.
  High intensity physical activity as for example running, playing football or tennis, measured in minutes (min.) pr week. Scale: 0 min, <30 min., 30-59 min., 60-120 min. and >120 min. Values <30 min. or 0 min. is considered low physical activity of high-intensity. 30-59 min. is considered medium physical activity of high intensity. Values > 60 min ia considered high physical activity level of high intensity.
  Low intensity physical activity as for example walking, doing the garden or cleaning the house, measured in minutes pr week. Scale: 0 min., <30 min., 30-60 min., 61-90 min., 91-150 min., 151-300 min. and >300 min. Values <60 min is considered low physical activity of low intensity. Values from 61-150 is considered medium physical activity of low intensity. Values from 151 or more is considered high physical activity level of low intensity.
Smoking measured by selfreported smoking status. A non-validated scale | Up to 7 years after stoma formation
  Exploration of the distribution of smoking in stoma patients with and without parastomal bulging. Smoking status is categorised as never smoked, stopped smoking for > 6 months, stopped smoking < 6 months, smoking occationally, smoking every day. The category never smoked will be categorised as 'never smoker'. The categories stopped smoking < or > than 6 months ago will be categorised as 'previous smoker'. The categories smoking occationally and smoking every day will be categorised as 'current smokers'.

CONTACTS AND LOCATIONS:
Locations (1):
- Marianne Krogsgaard, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No